CLINICAL TRIAL: NCT02507908
Title: '5-HIAA in Urine Versus 5-HIAA in Plasma in Patients With a Serotonin Producing Neuroendocrine Tumor'
Brief Title: 5-HIAA in Urine Versus 5-HIAA in Plasma Patients With a Serotonin Producing Neuroendocrine Tumor'
Acronym: 5-HIAA
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201500365
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumors; 5-hydroxyindolacetic acid; serotonin; isotope-dilution massa-spectrometer
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this observational laboratory study is to measure the correlation between 5-hydroxyindolacetic acid (5-HIAA) in platelet rich plasma and 5-HIAA in 24-hours urine collection in adult patients with a serotonin-producing neuro-endocrine tumor. Plasma and urine of included patients are collected and 5-HIAA values are measured with LCMS-MS and analysed.

DETAILED DESCRIPTION:
In midgut NETs serotonin production is most prominent. Patients with NETs producing excessive serotonin can develop carcinoid syndrome. Serotonin is a product of the 'tryptophan pathway'. Serotonin is metabolized in 5-hydroxyindolacetic acid (5-HIAA) and then excreted with urine. 5-HIAA in 24-hour urine collection is one of the parameters used for follow up in patients with a serotonin-producing neuroendocrine tumor. This measurement has some disadvantages; it could be stressful, the collection is not always precisely, furthermore the collection could be problematic, for example in patients with diarrhea.

Since October 2013 it is possible, because of a better measurement sensitivity, to measure reliably 5-HIAA in platelet rich plasma (PRP) by isotope-dilution massa-spectrometer (LCMS-MS). Recent publications show that 5-HIAA measured in PRP could have an additive value in diagnosis and follow up of patients with serotonin-producing NET.

Objective:

The primary objective is to measure the correlation between 5-HIAA in PRP and 5-HIAA in 24-hours urine collection in adult patients with a serotonin-producing neuro-endocrine tumor.

Secondary objective is to determine if increase or decrease of 5-HIAA in plasma is associated with disease progression.

Study design:

This is an observational laboratory study. Plasma and urine of included patients and collected in standard health care, are selected and the 5-HIAA's are measured with LCMS-MS. Also age, sex, diagnosis and clinical course of the patients will be collected from the medical record.

Study population:

In this study the investigators will use blood and urine of 60 patients with serotonin-producing neuro-endocrine tumors.

Main study parameters/endpoints:

The main endpoint of this study is the correlation between 5-HIAA in PRP and 5-HIAA in 24-hour urine collection. Secondary endpoint is the correlation between 5-HIAA in PRP and course of the disease, determined by CT-scan (if applicable).

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Serotonin in platelets > 5.4 nmol / 10^9 and 5-HIAA in 24-hours urine >3.8 mmol/mol creatinine
* Adult NET patients (aged ≥ 18 years of age)
* Blood and urine collection of the patient are collected within four days Patients are allowed to be included more than once.

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 Plasma and urine collections are used of adult patients with serotonin-producing neuro-endocrine tumors.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
the correlation between 5-HIAA in PRP and 5-HIAA in 24-hour urine collection | 4 days

SECONDARY OUTCOMES:
the course of the disease according to the course of 5-HIAA in plasma | 1 year
  the course of the disease according to the course of 5-HIAA in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Walenkamp, MDPhD, Principal Investigator — University Medical Centre
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands